CLINICAL TRIAL: NCT02771834
Title: Evaluation of the Association Between Osteoporosis and Postural Balance in Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Guilherme Carlos Brech, Phd, University of Sao Paulo
Other Study IDs: 320/09
Record Dates: First submitted 2016-05-10; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Postural Balance
Keywords: Postural balance; Osteoporosis; Postmenopause; Vitamin D; Kyfhosis; Muscle strength
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: women with osteoporosis
  Interventions: Other: Biomechanical analysis; Other: Kiphosis analysis; Other: Vitamin D level
- Control: women without osteoporosis
  Interventions: Other: Biomechanical analysis

INTERVENTIONS:
Other: Biomechanical analysis
Other: Kiphosis analysis
  Groups: Experimental
Other: Vitamin D level
  Groups: Experimental

SUMMARY:
The incidence of osteoporosis has been increasing, as have fractures resulting from falls.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate bipodal postural balance in postmenopausal women with and without lumbar osteoporosis. The specific objective is to determine the relationship between the degree of thoracic kyphosis and dosing of 25 OH vitamin D with postural balance in postmenopausal women with lumbar osteoporosis.

One hundred and twenty-six postmenopausal women between 55-65 years of age were evaluated and separated into two groups according to the bone mineral density values of their lumbar spine: the osteoporosis group and the control group.

Functional mobility was evaluated through the Timed Up and Go Test. Postural balance was evaluated using a AccuSway® model portable force platform, in standard standing position, with eyes open and closed, for 60". Data were collected, stored, and processed by the Balance Clinic® program, configured to 100 Hz frequency, with a frequency cut-off filter at 10 Hz.

Muscle strength was evaluated via a Biodex® isokinetic dynamometer in the concentric/concentric knee extension mode at 60o/s.

Dosing of 25 OH vitamin D and thoracic spine x-rays to determine the degree of kyphosis measured by the Cobb angle were performed in the osteoporosis group.

ELIGIBILITY:
Inclusion Criteria:

* absence of impairment of the vestibular, proprioceptive, auditory or neurological system, and/or any mental disturbances or disorders;
* no use of medications that might compromise postural balance;
* absence of lesions, surgery or disease that might have caused lower-limb joint limitations over the previous six months;
* absence of lower-limb dysmetria;
* presence of clinically normal gait, without claudication.

Exclusion Criteria:

* the presence of pain or inability to complete any of the tests
* along with occurrences of blood pressure increase before the strength evaluation.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 1 day

SECONDARY OUTCOMES:
Functional mobility | 1 day
  Was evaluated through the Timed Up and Go Test

OTHER OUTCOMES:
Postural balance | 1 day
  Was evaluated using a AccuSway® model portable force platform, in standard standing position, with eyes open and closed, for 60". Data were collected, stored, and processed by the Balance Clinic® program, configured to 100 Hz frequency, with a frequency cut-off filter at 10 Hz.
Muscle strength | 1 day
  Was evaluated via a Biodex® isokinetic dynamometer in the concentric/concentric knee extension mode at 60o/s.
Vitamin D level | 1 day
  Dosing of 25 OH vitamin D in a blood test
Degree of kyphosis | 1 day
  Thoracic spine x-rays to determine the degree of kyphosis measured by the Cobb angle were performed in the osteoporosis group

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brech GC, Ciolac EG, Peterson MD, Greve JM. Serum 25-hydroxyvitamin D levels are associated with functional capacity but not with postural balance in osteoporotic postmenopausal women. Clinics (Sao Paulo). 2017 Jan 1;72(1):11-16. doi: 10.6061/clinics/2017(01)03. PMID 28226027